CLINICAL TRIAL: NCT04702919
Title: Modifications Electrophysiologiques et de la Pulsatilité Cérébrale à la détection de Stimuli Nouveaux (Electro-PulCe)
Brief Title: Brain Changes in EEG and Brain Pulsatility to Novel Stimuli (Electro-PulCe)
Acronym: Electro-Pulce
Status: Completed | Type: Observational
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: RIPH3-RNI19 / Electro-Pulce; IdRCB (Other: 2020-A02170-39)
Record Dates: First submitted 2021-01-04; First posted 2021-01-11 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-02

CONDITIONS: Healthy Volunteers
Keywords: Brain Tissue Pulsatility (BTP); Electroencephalogram (EEG); Auditive oddball task; Tissue Pulsatility Imaging (TPI)

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy volunteers
  Interventions: Other: Registration; Other: Auditive oddball task

INTERVENTIONS:
Other: Registration — Synchronized recording of BTP in ultrasound, brain activity by EEG, heart rate and blood pressure.
Other: Auditive oddball task — Presentation of an auditory sequence, comprising 'Standard' (probability of occurrence: p = 0.90) and 'Deviants' (p = 0.10, targets) sounds via loudspeakers.

SUMMARY:
The oddball paradigm is one of the most widely used methods of brain exploration for the study of attentional processes. It allows the measurement, by means of an Electro-Enchephalogram (EEG), of evoked potentials reflecting the electrophysiological reactivity to the detection of novel stimuli within a stream of standard stimuli.

Other studies have recently suggested that, in addition to neuronal activation, certain other physiological processes related to cerebrovascular reactivity, such as the Brain Tissue Pulsatility (BTP), could also be sensitive to various cognitive processes and in particular to attentional processes.

In one of the latest studies published in collaboration with our group, it was shown that the amplitude of the electrophysiological response classically associated with attentional activity (P300 wave) was significantly correlated with the amplitude of BTP, suggesting the involvement of cerebrovascular processes in attentional functions. Nevertheless, in this study, the two methods of EEG and Tissue Pulsatility Imaging (TPI) were not synchronized, since TPI was performed at rest and not during the oddball task itself, and to date no study has sought to couple the methods of EEG and ultrasound TPI in an oddball paradigm, for a simultaneous characterization of neuronal and cerebrovascular responsiveness during attentional processes.

The general objective of this study will be to evaluate changes in BTP during the detection of novel stimuli in an oddball task in healthy volunteers, in which the two methods of TPI and EEG will be coupled and synchronized.

DETAILED DESCRIPTION:
The oddball paradigm is one of the most widely used methods of brain exploration for the study of attentional processes. It allows the measurement, by means of an Electro-Enchephalogram (EEG), of evoked potentials reflecting the electrophysiological reactivity to the detection of novel stimuli within a stream of standard stimuli. Numerous studies have thus used the oddball paradigm to identify the neuronal reactivity involved in attentional orientation towards target stimuli.

Other studies have recently suggested that, in addition to neuronal activation, certain other physiological processes related to cerebrovascular reactivity, such as the Brain Tissue Pulsatility (BTP), could also be sensitive to various cognitive processes and in particular to attentional processes. Ultrasound measurement of BTP is made possible by recent advances in both the development of ultrasound equipment and ultrasound signal processing. Our team and others have validated the measurement of BTP by ultrasound (Tissue Pulsatility Imaging - TPI) in healthy volunteers and clinical populations, and our results suggest that the mechanisms of BTP are significantly influenced by cerebrovascular physiology.

In one of the latest studies published in collaboration with our group, it was shown that the amplitude of the electrophysiological response classically associated with attentional activity (P300 wave) was significantly correlated with the amplitude of BTP, suggesting the involvement of cerebrovascular processes in attentional functions. Nevertheless, in this study, the two methods of EEG and TPI were not synchronized, since TPI was performed at rest and not during the oddball task itself, and to date no study has sought to couple the methods of EEG and ultrasound TPI in an oddball paradigm, for a simultaneous characterization of neuronal and cerebrovascular responsiveness during attentional processes.

The general objective of this study will be to evaluate changes in BTP during the detection of novel stimuli in an oddball task in healthy volunteers, in which the two methods of TPI and EEG will be coupled and synchronized.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 45 years old included
* Normal hearing

Exclusion Criteria:

* History of neurologic, psychiatric or cardiologic diseases (stroke, severe head trauma, mood disorder, psychotic disorder, coronary syndrome, heart rhythm disorder, etc.)
* Treatment which could impact Brain Tissue Pulsatility (Beta-Blockers, Neuroleptics, etc...) and electrophysiological (Sedatives, Benzodiazepines, etc...) parameters.
* Legal protection measures
* Opposition to data processing

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy volunteer
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2022-02-21 (Actual); Primary Completion 2022-06-17 (Actual); Study Completion 2022-06-17 (Actual)

PRIMARY OUTCOMES:
Change in Brain Tissue Pulsatility indexes | Baseline and during the auditive oddball task (20 minutes)
  Measured by the Tissue Pulsatility Imaging technique - TPI

SECONDARY OUTCOMES:
P300 wave | Baseline and during the auditive oddball task (20 minutes)
  Evoked potential P300 measured by Electroencephalogram (EEG)
Heart Rate changes and Heart Rate Variability | Baseline and during the auditive oddball task (20 minutes)
  Measured by electrocardiogram (ECG)
Arterial pressure blood | Baseline and during the auditive oddball task (20 minutes)
  Measured by a non-invasive and continuous blood pressure bracelet.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Desmidt, Md-PhD, Principal Investigator — University Hospital, Tours
Locations (1):
- Paedopsychiatry department, University Hospital, Tours, Tours, France